CLINICAL TRIAL: NCT00894478
Title: Improving Lesion Detection in Children With MRI-negative Partial Epilepsy Using Diffusion Tensor Imaging
Brief Title: Improving Lesion Detection in Children With Magnetic Resonance Imaging (MRI)-Negative Partial Epilepsy Using Diffusion Tensor Imaging
Status: Completed | Type: Observational
Sponsor: The Hospital for Sick Children (Other)
Responsible Party: Principal Investigator, Elysa Widjaja, Staff Neuroradiologist, The Hospital for Sick Children
Other Study IDs: 1000013137
Record Dates: First submitted 2009-05-06; First posted 2009-05-07 (Estimated); Last update posted 2013-09-10 (Estimated); Status verified 2013-09

CONDITIONS: Localization-related Epilepsy; Partial Epilepsy
Keywords: MRI-Negative; Diffusion tensor imaging; Localization-related epilepsy; Partial Epilepsy; Children
MeSH Terms: conditions — Epilepsies, Partial | interventions — Diffusion Tensor Imaging; Magnetoencephalography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- 1: 12 children with MRI-negative partial epilepsy who are being worked-up for epilepsy surgery
  Interventions: Procedure: Diffusion Tensor Imaging (DTI); Procedure: Magnetoencephalography
- 2: 12 children with MRI-visible FCD who are being worked-up for epilepsy surgery
  Interventions: Procedure: Diffusion Tensor Imaging (DTI); Procedure: Magnetoencephalography
- 3: Control Group- Healthy Volunteers
  Interventions: Procedure: Diffusion Tensor Imaging (DTI)

INTERVENTIONS:
Procedure: Diffusion Tensor Imaging (DTI) — MR and DTI: MRI and DTI will be done using 3.0T Philips MR scanner (Philips Medical Systems, Best, The Netherlands) using an eight channel head coil. DTI and axial 3D T1 will be performed on patients and controls.
  1. DTI will be performed using single shot diffusion-weighted echo planar imaging, b=1000s/mm2 and 15 noncollinear directions (TR/TE=10,000/60 ms, slice thickness=2mm, field of view=22cm, matrix=112x112, NEX=2)
  2. Axial 3D T1 (TR/TE=4.9/2.3 ms, slice thickness=1 mm, field of view = 24 cm, matrix=220x220, NEX=1) Patients will have additional sequences (axial and coronal T2, proton density and FLAIR) as part of their clinical scan
Procedure: Magnetoencephalography — MEG will be performed using a whole-head Omega 151-channel gradiometer system (VSM MedTech, Port Coquitalam, BC, Canada). At least 15 2-minute periods of spontaneous data will be recorded with a sampling rate for data acquisition of 625Hz, a bandpass filter of 10 to 70 Hz and a notch filter of 60 Hz.
  Other Names: MEG
  Groups: 1; 2

SUMMARY:
Focal cortical dysplasia is one of the most common lesions responsible for medically refractory epilepsy in the pediatric population. In patients with medically intractable epilepsy, surgery is the only treatment that will lead to seizure freedom. The outcome of epilepsy surgery is worse in patients when there is no lesion identified on routine structural MRI, also known as MRI-negative partial epilepsy. Diffusion tensor imaging (DTI), a novel MRI technique, can be used to evaluate the integrity of the microstructure of the white matter, even when the white matter appears normal on routine MRI.

DETAILED DESCRIPTION:
The aims of this study are firstly to identify DTI abnormalities in the white matter of children with MRI-negative partial epilepsy and MRI-visible FCD compared to normal controls; and secondly to determine if the location of DTI identified abnormalities correlate with the epileptogenic zone as defined using magnetoencephalography (MEG) dipole clusters. Our hypotheses are firstly DTI can demonstrate the anatomic delineation of white matter abnormalities in MRI-negative partial epilepsy and the alteration in DTI indices are similar in MRI-negative partial epilepsy and MRI-visible FCD, which is the positive control; and secondly the anatomical location of DTI identified abnormalities correlate with the epileptogenic zone as defined by MEG dipole clusters. The long-term goal of this study is to improve detection of subtle lesions in children with MRI-negative partial epilepsy so as to improve the surgical outcome of these patients who undergo epilepsy surgery for seizure control.

ELIGIBILITY:
Inclusion Criteria:

MRI negative partial epilepsy group:

* Patients diagnosed with partial epilepsy according to the International League Against Epilepsy (ILAE) standard [53]
* MRI study reported as normal
* Age ranging from 6-18 years (DTI indices alter with myelination and the changes are most marked from birth to 4 years of age)

MRI-visible FCD group:

* Patients diagnosed with partial epilepsy according to the ILAE standard [53]
* Visual assessment of MRI demonstrates one or more features of FCD

  * Cortical thickening
  * Alteration in sulci and gyri pattern, including deep sulci
  * Blurring of gray-white matter transition
  * T2 signal prolongation of the cortex and subcortical white matter
  * High T1 signal in the cortex
* Age ranging from 6-18 years (DTI indices alter with myelination and the changes are most marked from birth to 4 years of age)

Normal controls:

* Subjects with no history of neurological diseases
* Age ranging from 6-18 years (most children under the age of 6 years are unable to tolerate the MR examination without general anesthesia or sedation).
* No requirement of general anesthesia or sedation

Exclusion Criteria:

* Subjects with contraindications for MR imaging (i.e. retained foreign bodies, implants)
* Subjects with claustrophobia
* Controls with a prior history of traumatic brain injury, neurological disorder, cerebral palsy, developmental delay or learning disability
* Controls who require general anesthesia or sedation

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Patients will be identified from the epilepsy clinic and seizure rounds and who have had previous MRI in an outside institution or prior MRI at least two years ago at the Hospital for Sick Children.
  Control children will be recruited through hospital publications and from families participating in the study (healthy siblings)
Sampling Method: Non-Probability Sample
Enrollment: 64 (Actual)
Dates: Start 2009-05; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Identify DTI changes in the white matter of children with MRI-negative partial epilepsy and MRI-visible FCD using voxel-by-voxel analysis of FA and MD maps compared to normal controls. | 1 timepoint; immediately after MRI/DTI

SECONDARY OUTCOMES:
Determine if the lobar location of abnormal FA and MD correlate with the lobar location of MEG defined epileptogenic zone in MRI-negative partial epilepsy and MRI-visible FCD. | 1 timepoint; immediately after MRI/DTI

CONTACTS AND LOCATIONS:
Overall Officials: Elysa Widjaja, MD, Principal Investigator — The Hospital for Sick Children
Locations (1):
- The Hospital for Sick Children, Toronto, Ontario, Canada